CLINICAL TRIAL: NCT01599182
Title: Metabolic Effects of Treatment in Intermediate and High-Risk Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: Grand River Regional Cancer Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 17074; 2011-0454 (Other: Tri-Hospital Research Ethics Board)
Record Dates: First submitted 2012-02-20; First posted 2012-05-15 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Measurements related to glucose, lipid and immune metabolism will be measured.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High-Risk Prostate Cancer
- Intermediate-Risk Prostate Cancer

SUMMARY:
This study will work towards understanding the changes in your body (metabolism) that develop with treatment in prostate cancer. Hormonal therapies such as ADT often result in detrimental changes in body composition, including lean tissue loss and fat gains, compared to those patients receiving radiation therapy. These changes in body composition are linked to risk of diabetes and cardiovascular disease in survivorship. The investigators will be evaluating 50 patients to primarily examine the changes in metabolism, nutrition, physical function and body composition at the end of treatment, 6 weeks and 6 months following the end of treatment. Patients will continue to be followed every 6 months for up to 5 years following the end of treatment. The investigators findings will provide a new perspective for future work and novel approaches in the treatment of prostate cancer.

DETAILED DESCRIPTION:
Intermediate and high risk prostate cancer patients generally undergo either watchful waiting, surgery, RT alone or RT in conjunction with androgen deprivation therapy (ADT). Prostate cancer patients who receive upfront ADT exhibit drastic reductions in testosterone, resulting in the loss of a key anabolic signal and ultimately muscle loss and adipose tissue gain. In non-malignant populations, these changes in body composition are associated with the development of insulin resistance and metabolic syndrome. Hypogonadism is also independently predictive of hyperinsulinemia and metabolic syndrome, and may be the consequence of ADT, increased saturated fat intake, inactivity as well as unhealthy changes in body composition during the treatment time-course. However, it is thought that obesity itself is associated with atherogenic profiles, insulin resistance, biochemical failure, increased risk of cancer recurrence and/or metabolic syndrome in prostate cancer. The loss of muscle is largely attributed to reduced anabolic stimulus due to inactivity and reduced androgen hormones from ADT. As skeletal muscle has an important role in glucose disposal, using RT alone does not reduce androgen hormone levels and may maintain muscle mass to prevent the deleterious metabolic effects exhibited with ADT. Thus, different forms of therapy may present with diverse changes in body composition and ultimately metabolic implications.

While there are discrepancies in the success of ADT therapy, this form of therapy invariably results in several detrimental metabolic changes that predispose prostate cancer patients and survivors to developing chronic diseases such as diabetes and cardiovascular disease as well as a greater risk of cancer recurrence. In fact, prostate cancer patients who undergo radical prostatectomy and androgen deprivation therapy, not only lose muscle mass while undergoing treatment but also develop a greater risk of mortality from cardiovascular disease as compared to prostate cancer patients receiving other forms of therapy. To date, no studies have examined the metabolic effects that develop with ADT and/or radiation therapy. The results of the proposed study will indicate the potential metabolic changes that develop with therapy. It is important to identify these unhealthy changes early so that specific nutrition and exercise protocols may be used to improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate or high risk prostate cancer patients who have >T2a or Gleason >6 or PSA >10
* Able to communicate in English
* Have sufficient cognitive ability to participate and provide informed consent

Exclusion Criteria:

* Any known diagnosis of cardiovascular disease, diabetes, HIV, uncompensated thyroid disease
* Pre-existing injuries or health conditions that prevents the patient's participation in exercise
* Any previous diagnosis of cancer or anti-neoplastic treatment (other than melanoma skin cancer) which is not in remission for at least 3 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intermediate and high risk prostate cancer patients with >T2a or Gleason > 6 or PSA >10 would be offered participation in this study.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Glucose Metabolism | Baseline, 7 weeks, 30 weeks
  Oral glucose tolerance tests will be performed at each time point to assess changes in the body's ability to metabolize glucose. As such, other related parameters such as insulin and c-peptide will be measured to understand potential changes in glucose over the indicated time frame. As this is an observational study, safety issues are not anticipated. However, abnormal measures of glucose and insulin will be reported to a given participant's family physician.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Mourtzakis, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada